CLINICAL TRIAL: NCT01811563
Title: Clinical and Functional Outcomes Following Total Knee Replacement Using Two Different Implants
Brief Title: Total Knee Arthroplasty: Functional and Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00043737; 193447 (Other Grant/Funding Number: Stryker)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Replacement; Lower Quarter Y-Balance Test; Functional Outcomes; Patient Reported Outcomes
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stryker (Active Comparator): Subjects will be receiving the Stryker Triathlon total knee replacement
  Interventions: Device: Stryker
- Zimmer (Active Comparator): Subjects will be receiving a Zimmer NexGen total knee replacement
  Interventions: Device: Zimmer

INTERVENTIONS:
Device: Zimmer
  Arms: Zimmer
Device: Stryker
  Arms: Stryker

SUMMARY:
The purpose of this study is to assess the differences in functional and patient reported outcomes between total knee replacement (TKA) implants. In addition, this work will examine the correlation between functional assessments and patient reported outcomes following surgery. All subjects will complete assessments preoperatively, 4-6 weeks following TKA and then one year following TKA. Subjects will complete a series of patient reported outcomes as well as a series of functional outcomes at each of the time points of interest. The analysis will include a repeated measures design to determine differences between groups across time as well as correlations between the functional and patient reported outcomes. This work will hopefully determine the importance of using objective functional outcomes following TKA as well as determining the need for patient assessments out to one year following surgery.

DETAILED DESCRIPTION:
The number differences in subjects analyzed from baseline to 6 weeks to 52 weeks are due to the fact that we did not use the 6 week time point in the final analysis based on the clinical decision that 6 weeks was too early in recovery to provide accurate information for clinical decision making. Therefore the patients used in the final analysis were those subjects who were able to and completed the assessment at pre-op and 1 year post-op which is how we get to the 20 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring primary total knee replacement
2. Patients willing and able to comply with the follow-up visits and evaluations
3. Patients willing to sign informed consent approved by the Institutional Review Board

Exclusion Criteria:

1. Patients with inflammatory arthritis
2. Patients with diabetic neuropathy
3. Patients unable to ambulate without the use of an assistive device prior to surgery
4. Patients unable to stand in single limb stance on each foot prior to surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel S Wellman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients signed consent form but 12 were withdrawn at the time of surgery because they required a different implant not included in the study.
Groups:
- Stryker: Subjects will be receiving the Stryker Triathlon total knee replacement
  Stryker
- Zimmer: Subjects will be receiving a Zimmer NexGen total knee replacement
  Zimmer
Period: Overall Study
Arm/Group | Stryker | Zimmer
Started | 25 | 23
Completed | 20 | 20
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 2
Not completed — Incorrect Randomization procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stryker | Zimmer | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.0) | 63.1 (7.3) | 62.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Quarter Y-Balance Test (YBT-LQ) (Dynamic Balance) From Baseline to 6 Weeks Following Total Knee Replacement
Description: The lower quarter y-balance test (YBT-LQ) is a test of dynamic balance in unilateral stance that has been deemed to be reliable and valid. The YBT-LQ consists of each patient standing on one leg and reaching as far as they can with their non-stance leg in the anterior, posteromedial and posterolateral direction while standing on the other foot on a centralized stance platform. The composite score is calculated as the sum of the three reach directions divided by 3 time the limb length and will be reported as a percentage of limb length.
Time Frame: Baseline (Pre-Operative) to 6 weeks following total knee replacement
Population: Only subjects that were able to complete all of the YBT assessments at 6 weeks post total knee replacement were included in the analyses.
Measure: Mean (Standard Deviation); unit: % of limb length
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 21 | 22
% of limb length
  YBT-LQ Composite Pre-Operative | 69.98 (8.18) | 67.52 (12.22)
  YBT-LQ Composite 6 weeks | 73.25 (7.95) | 73.32 (9.15)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for implant independent of time; p = 0.661, ANOVA
Statistical Analysis 2: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for time independent of implant; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Stryker vs Zimmer; Test type: Equivalence — Interaction between implant and time; p = 0.270, ANOVA

2. Primary Outcome: Change in Lower Quarter Y-Balance Test (YBT-LQ) (Dynamic Balance) From Baseline to 52 Weeks Following Total Knee Replacement
Description: as for outcome 1
Time Frame: Baseline (Pre-Operative) to 52 weeks following total knee replacement
Population: Subjects used in the final analysis were those subjects who completed the assessment at pre-op and 1 year post-op (20 subjects per arm).
Measure: Mean (Standard Deviation); unit: % of limb length
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 20 | 20
% of limb length
  YBT-LQ Composite Pre-Operative | 79.45 (10.46) | 79.24 (7.89)
  YBT-LQ Composite Post-Op 52 Weeks | 70.44 (9.31) | 69.42 (13.39)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for implant independent of time; p = 0.856, ANOVA; Main effect for implant, LQ-YBT Baseline to 52 weeks
Statistical Analysis 2: Comparison: Stryker vs Zimmer; Test type: Equivalence — Time independent of implant, Baseline to 52 Weeks; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Stryker vs Zimmer; Test type: Equivalence — Implant by Time interaction, Baseline to 52 Weeks between Zimmer and Stryker; p = 0.822, ANOVA

3. Secondary Outcome: Change in Walking Speed From Baseline to 52 Weeks Following Total Knee Replacement.
Description: Each subject will complete three walking trials at a self-selected comfortable walking speed along a 5 meter walkway in order to record walking speed at each time point.
Time Frame: Baseline and 52 weeks following total knee replacement
Measure: Mean (Standard Deviation); unit: miles per hour
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 20 | 20
miles per hour
  Walking Speed Pre-Operative | 1.22 (0.21) | 1.16 (0.28)
  Walking Speed Post-Op 52 Weeks | 1.41 (0.23) | 1.28 (0.23)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for implant, Baseline to 52 weeks; p = .158, ANOVA
Statistical Analysis 2: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for time, Baseline to 52 weeks; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Stryker vs Zimmer; Test type: Equivalence — Interaction of time by implant, Baseline to 52 weeks; p = 0.365, ANOVA

4. Secondary Outcome: Walking Speed at 6 Weeks Following Total Knee Replacement.
Description: as for outcome 3
Time Frame: 6 weeks following total knee replacement
Measure: Mean (Standard Deviation); unit: miles per hour
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 25 | 23
miles per hour | 1.21 (0.28) | 1.19 (0.22)

5. Other Pre Specified Outcome: Change in University of California, Los Angeles (UCLA) Activity Score From Baseline to 52 Weeks Following Total Knee Replacement.
Description: The UCLA activity score is a validated patient reported outcome of overall physical activity. Results on a scale of 1 to 10, 1 is "Wholly Inactive, dependent on others, and can not leave residence" and 10 is "Regularly participates in impact sports".
Time Frame: Baseline and 52 weeks following total knee replacement
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 20 | 20
units on a scale
  UCLA Activity Pre-Operative | 4.19 (1.33) | 3.83 (1.38)
  UCLA Activity Post-Op 52 Weeks | 5.90 (1.55) | 5.61 (1.91)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for implant, baseline to 52 weeks; p = .416, ANOVA
Statistical Analysis 2: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect for time, Baseline to 52 weeks; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Stryker vs Zimmer; Test type: Equivalence — Implant by time interaction, baseline to 52 weeks; p = 0.917, ANOVA

6. Other Pre Specified Outcome: University of California, Los Angeles (UCLA) Activity Score at 6 Weeks Following Total Knee Replacement.
Description: as for outcome 5
Time Frame: 6 weeks following total knee replacement
Population: Only subjects who were able to complete the UCLA at six weeks were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 25 | 22
units on a scale | 4.48 (1.42) | 4.73 (1.52)

7. Other Pre Specified Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Total From Baseline to 52 Weeks Following Total Knee Replacement.
Description: The KOOS is a standardized and validated patient outcome score that assesses functional limitation in patient with knee problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: Baseline (Pre-Operative) and 52 weeks following total knee replacement
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 20 | 20
units on a scale
  KOOS Total, Baseline Pre-Operative | 45.60 (12.32) | 46.08 (13.50)
  KOOS Total, Post-Op 52 week | 67.32 (35.62) | 64.24 (38.79)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect by implant, Baseline to 52 weeks; p = 0.830, ANOVA
Statistical Analysis 2: Comparison: Stryker vs Zimmer; Test type: Equivalence — Main effect by time, baseline to 52 weeks; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Stryker vs Zimmer; Test type: Equivalence — Interaction between implant and time, baseline to 52 weeks; p = 0.728, ANOVA

8. Other Pre Specified Outcome: Change in Forgotten Joint Score (FJS) From 6 Weeks to 52 Weeks Following Total Knee Replacement.
Description: The FJS is a patient reported measure of how bothersome the total joint replacement is for them, how much it affects daily activity and how much they are aware of the implant. The FJS is a 12-question survey regarding functional outcome, pain, stability, daily living, activity and sport. Scoring is from 0 to 4 with 0 as the best outcome; a low score means high satisfaction. Not all questions must be answered to score, all responses are summed and the total is divided by number of completed items multiplied by 25, with the final result subtracted from 100. The score range is from 0 to 100 with the highest score of 100 indicating the best outcome (the joint is completely "forgotten") and 0 indicating the worst outcome.
Time Frame: 6 weeks and 52 weeks following total knee replacement
Population: Participants who completed the Forgotten Joint Score (FJS) at week 6 and week 52. Not all subjects completed the FJS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 20 | 20
units on a scale
  FJS, at 6 weeks: number analyzed (Participants) | 19 | 17
  FJS, at 6 weeks | 69.63 (20.9) | 76.59 (20.39)
  FJS, at 52 weeks | 37.7 (21.4) | 30.8 (29.6)
Statistical Analysis 1: Comparison: Stryker vs Zimmer; Test type: Equivalence — Between implants at 6 weeks; p = 0.319, t-test, 2 sided

9. Other Pre Specified Outcome: Knee Society Score (KSS)
Description: The KSS is a patient reported measure of knee function that is specific to patients who are scheduled to receive or have previously had a total knee replacement. This outcome measures both patient reported pain and function changes from prior to surgery through recovery. The score range is from 0 to 100. The highest score of 100 points will be obtained by a well-aligned knee with no pain, 125 degrees of motion, and negligible anteroposterior and mediolateral instability.
Time Frame: Baseline (Pre-Operative), 6 weeks and 52 weeks following total knee replacement
Population: Only 20 subjects in each arm completed the assessment at 1 year post-op.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 25 | 23
units on a scale
  KSS Satisfaction, Baseline Pre-Operatively | 11.1 (5.2) | 13.6 (8.8)
  KSS Satsifaction, 6 weeks | 28.9 (7.3) | 29.5 (8.8)
  KSS Functional Activity, Baseline | 44.3 (11.2) | 47.0 (13.7)
  KSS Functional Activity, 6 weeks | 60.8 (18.1) | 61.6 (16.7)
  KSS Functional Activity, 52 weeks Post-operative: number analyzed (Participants) | 20 | 20
  KSS Functional Activity, 52 weeks Post-operative | 67.3 (35.6) | 64.2 (38.8)

10. Other Pre Specified Outcome: Sit to Stand Time
Description: The sit to stand test requires patients to stand up and sit down as many times as possible in 10 seconds from a standard arm chair.
Time Frame: Baseline (Pre-Operative), 6 weeks and 52 weeks following total knee replacement
Population: The 6 week time point was not used in the final analysis based on the clinical decision that 6 weeks was too early in recovery to provide accurate information for clinical decision making. Subjects used in the final analysis were those subjects who completed the assessment at pre-op and 1 year post-op (20 subjects per arm).
Measure: Mean (Standard Deviation); unit: Number of times
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 25 | 23
Number of times
  Sit to stand Pre-Operative | 3.90 (0.95) | 4.34 (1.34)
  Sit to stand Post-Op 6 weeks | 4.5 (1.7) | 4.6 (1.1)
  Sit to stand Post-Op 52 weeks: number analyzed (Participants) | 20 | 20
  Sit to stand Post-Op 52 weeks | 5.40 (1.45) | 5.47 (1.81)

11. Other Pre Specified Outcome: Timed Get up and go
Description: The timed up and go requires a patient to rise from a chair walk three meters around a piece of tape and return to the chair again as quickly as possible.
Time Frame: Baseline (Pre-Operative), 6 weeks and 52 weeks following total knee replacement
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Stryker | Zimmer
Number analyzed (Participants) | 24 | 23
Seconds
  Timed up and go Pre-Operative | 9.55 (3.86) | 9.07 (2.48)
  Timed up and go Post-Op 6 weeks | 9.38 (3.58) | 8.89 (1.89)
  Timed up and go Post-Op 52 weeks: number analyzed (Participants) | 20 | 20
  Timed up and go Post-Op 52 weeks | 6.99 (1.8) | 7.17 (1.39)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Stryker | Zimmer
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 1/25 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stryker (N=25) | Zimmer (N=23)
Patient fell while completeing the 6 weeks testing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient was being tested at the 6 week post-op time point in the clinic and was asked to complete the single leg stance test as part of the functional assessments that were to be completed at this study visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No